CLINICAL TRIAL: NCT06217042
Title: HR070803 in Combination With Oxaliplatin, 5-fluorouracil, Calcium Folinate Versus Gemcitabine in Combination With Capecitabine as Adjuvant Therapy for Pancreatic Cancer: an Open, Randomized, Multicenter Phase III Trial.
Brief Title: HR070803 in Combination With Oxaliplatin, 5-fluorouracil/LV Versus GX as Adjuvant Therapy for Pancreatic Cancer
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xian-Jun Yu, Professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HR070803-307
Record Dates: First submitted 2024-01-10; First posted 2024-01-22 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Oxaliplatin; Fluorouracil; Leucovorin; Gemcitabine; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HR070803+Oxaliplatin+5-FU/LV (Experimental): HR070803; Oxaliplatin; 5Fluorouracil; Calcium folinate
  Interventions: Drug: HR070803; Oxaliplatin; 5Fluorouracil; Calcium folinate
- GX (Active Comparator): gemcitabine; capecitabine
  Interventions: Drug: gemcitabine; capecitabine

INTERVENTIONS:
Drug: HR070803; Oxaliplatin; 5Fluorouracil; Calcium folinate — Oxaliplatin 85 mg/m² D1 over 2 hours, followed by HR070803 60 mg/m² D1 over 90 minutes, after the Folinic acid infusion is started. Folinic acid 400 mg/m² D1, IV infusion over 1 hours. 5-FU 2400 mg/m² D1 IV continuous infusion over 46 hours.
  These drugs are given once every 2 weeks, 12 cycles, 24 weeks.
  Arms: HR070803+Oxaliplatin+5-FU/LV
Drug: gemcitabine; capecitabine — Gemcitabine 1000mg/m² is given as an i.v. infusion over 30 minutes, administered on day 1, 8 and 15 out of 28 days. Capecitabine 1660mg/m²/day in two divided doses administered orally for 21 days followed by 7 days'rest .
  Arms: GX

SUMMARY:
The purpose of this study is to look at the efficacy and safety of HR070803 in combination with 5 fluorouracil/leucovorin (5FU/LV) plus oxaliplatin compared to gemcitabine + capecitabine treatment as adjuvant therapy in patients with resected pancreatic cancer.

DETAILED DESCRIPTION:
STUDY DESIGN/ Evaluation criteria Main criterion: efficacy. The main criterion is the disease-free survival. Disease-free survival is defined as the time from date of randomization until the date of the first cancer-related event, second cancer, or death from any cause. Patients without event at the time of analysis will be censored at the date of last follow-up visit.

Secondary criteria include Overall survival. OS is defined as the time from date of randomization until the date of death from any cause. Patients who are still living at the time of analysis will be censored at the date of last follow-up visit.

Secondary criteria also include 3-year disease-free survival rate/overall survival rate and 5-year disease-free survival rate/overall survival rate.

Tolerance Patients evaluable for toxicity must have received one investigational drug.

ELIGIBILITY:
Inclusion Criteria:

1. ECOG performance status 0 or 1
2. Histologically confirmed resected ductal pancreatic adenocarcinoma with macroscopic complete resection (R0 and R1).
3. Life expectancy of greater than or equal to 6 months.
4. Full recovery from surgery and patient is scheduled to start treatment within 3 weeks to 12 weeks after surgery.
5. Acceptable hematology parameters and blood chemistry levels.
6. Able and willing to provide a written informed consent.

Exclusion Criteria:

1. Patients with pancreatic cancer originating from extrapancreatic ductal epithelium, including pancreatic neuroendocrine carcinoma, acinar cell carcinoma of the pancreas, pancreatoblastoma, and solid-pseudopapillary tumor;
2. Presence of or history of metastatic or locally recurrent pancreatic adenocarcinoma.
3. CA 19-9> 180 U / ml within 21 days of registration on study.
4. Prior neo-adjuvant treatment, radiation therapy, or systemic therapy for pancreatic adenocarcinoma.
5. Severe infection (> CTCAE grade 2), such as severe pneumonia, bacteremia, infection complications, etc. requiring inpatient treatment, occurred within four weeks before enrollment, and symptoms and signs of infection requiring intravenous antibiotic therapy (except for prophylactic antibiotics) occurred within two weeks before enrollment;
6. Patients with cardiac clinical symptoms or diseases that are not well controlled, such as: (1) Patients with NYHA class 2 and above cardiac failure; (2) unstable angina; (3) myocardial infarction that occurred within 6 months; (4) clinically significant supraventricular or ventricular arrhythmia requiring treatment or intervention.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 524 (Estimated)
Dates: Start 2024-02-05 (Estimated); Primary Completion 2027-03-30 (Estimated); Study Completion 2028-07-30 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival (DFS) | From study start until 338 DFS events have occurred (approximately 21 months after last patient enrollment)
  Disease-free survival is defined as the time from date of randomization until the date of the first cancer-related event, second cancer, or death from any cause.

SECONDARY OUTCOMES:
Overall survival (OS) | From date of randomization until the date of death from any cause, assessed up to 37 months
  OS is defined as the time from date of randomization until the date of death from any cause.
3-year disease-free survival rate | up to 36 months following the date the first patient was randomized
  Disease-free survival within 3 years
5-year disease-free survival rate | up to 60 months following the date the first patient was randomized
  Disease-free survival within 5 years
3-year overall survival rate | up to 36 months following the date the first patient was randomized
  Overall survival within 3 years
5-year overall survival rate | up to 60 months following the date the first patient was randomized
  Overall survival within 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Si Shi, PhD, Principal Investigator — Fudan University
Locations (1):
- Department of Pancreatic Surgery, Fudan University Shanghai Cancer Center; Pancreatic Cancer Institute, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
study protocol and ICF, CSR will be shared.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Ending of trials, preserved for 10 years.
Access Criteria: Researchers within pancreatic cancer field.